CLINICAL TRIAL: NCT05974436
Title: Green Dialysis: Hemodialysis With Reduced Dialysate Flow
Brief Title: Green Dialysis: Dialysis With Reduced Dialysate Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2023-0170
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Uremic Syndrome
Keywords: dialysis efficiency; lowered dialysis fluid
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hemodiafiltration with high-flux dialyzer (Experimental): Patients are dialysed at midweek using hemodiafiltration (autoflow) with an FX800 Cordiax high-flux dialyzer, with dialysate flow of 700mL/min
  Interventions: Other: Blood and dialysate sampling
- Hemodialysis with medium cut-off dialyzer and high dialysate flow (Experimental): Patients are dialysed at midweek using hemodialysis with a Theranova 400 medium cut-off dialyzer with dialysate flow of 700mL/min
  Interventions: Other: Blood and dialysate sampling
- Hemodialysis with medium cut-off dialyzer and low dialysate flow (Experimental): Patients are dialysed at midweek using hemodialysis with a Theranova 400 medium cut-off dialyzer with dialysate flow of 300mL/min
  Interventions: Other: Blood and dialysate sampling

INTERVENTIONS:
Other: Blood and dialysate sampling — Blood is sampled from the inlet and outlet dialyzer bloodline at 5min after dialysis start.
  Spent dialysate is sampled from the outlet dialysate line at 5, 30, 90 and 240min after dialysis start.
  Blood and dialysate samples are analysed for different uremic toxins. Dialysis efficiency is calculated from the analysed toxin concentrations.

SUMMARY:
Hemodialysis patients consume per year 18.720-26.208L of dialysis fluid (i.e. water). From an ecological point of view, the present study investigated whether reducing this water amount has an impact on the extraction and total solute removal of different uremic toxins. The efficiency of hemodiafiltration with a standard high-flux dialyzer is compared to hemodialysis with a medium cut-off dialyzer with a dialysate flow of either 700mL/min or 300mL/min.

DETAILED DESCRIPTION:
Hemodialysis is currently performed with dialysate flows in the range 500 and 700mL/min respectively in hemodialysis and hemodiafiltration mode. With a standard daytime dialysis scheme of three times four hours a week, each patient consumes up to 360-504L dialysate per week or 18.720-26.208L per year.

From an ecological point of view, one can wonder whether patients can be dialyzed adequately enough using hemodialysis mode with a lower dialysate flow, and as such consuming less water.

Changing the mode from hemodiafiltration to hemodialysis mainly has an impact on the removal of larger toxins which benefit of the convective transport. Lowering dialysate flow in hemodialysis mode mainly has an impact on the removal of small water soluble toxins which are mainly removed by diffusion. For this transport, different parameters are important: blood and dialysate flow, dimensions of the membrane (surface area and thickness), fiber diameter, and extra-luminal space, and membrane porosity (Sieving coefficient). This also implies that, for the same blood and dialysate flow, the choice of the dialyzer will determine toxin transport. The use of a medium cut-off membrane with smaller and more open fibers might thus be more adequate in hemodialysis mode than a standard high-flux dialyzer with wider fibers.

The aim of this study is to quantify instant extraction and overall total solute removal of representative uremic toxins in hemodiafiltration with a standard high-flux hemodialyzer versus hemodialysis with a medium cut-off membrane, either with a standard or reduced dialysate flow.

ELIGIBILITY:
Inclusion Criteria:

* stable chronic hemodialysis patient
* well functioning vascular access

Exclusion Criteria:

* active infection
* malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Dialysis efficiency | three midweek dialysis sessions (3 arms)
  Dialyzer extraction and total solute removal are measured and calculated for different uremic toxins

CONTACTS AND LOCATIONS:
Overall Officials: Van Biesen, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium